CLINICAL TRIAL: NCT00279721
Title: Phase II Study of Intensity-modulated Radiation (IMRT)With Simultaneous Integrated Boost (SIB) as Adjuvant Treatment for High Risk Resected Well-differentiated Thyroid Cancer.
Brief Title: Phase II Study of IMRT With SIB as Adjuvant Treatment for High Risk Resected Well-differentiated Thyroid Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alberta Health services (Other)
Organization: AHS Cancer Control Alberta (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18916
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2011-07

CONDITIONS: Thyroid Neoplasms
Keywords: thyroid neoplasms; intensity modulated radiation; radiotherapy
MeSH Terms: conditions — Thyroid Neoplasms

INTERVENTIONS:
Procedure: IMRT

SUMMARY:
Resected well-differentiated thyroid neoplasms with at least one high risk feature will receive adjuvant radiation using IMRT with SIB. The acute toxicity and locoregional control rate at 2 years will be recorded.

DETAILED DESCRIPTION:
Resected well-differentiated thyroid neoplasms with at least one high risk feature will receive adjuvant radiation using IMRT with SIB. The acute toxicity and locoregional control rate at 2 years will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* resected well-differentiated throid cancer with at least one high risk feature for locoregional recurrence

Exclusion Criteria:

* medullary or anaplastic thyroid cancer, unresectable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
toxicity according to RTOG criteria
locoregional control

CONTACTS AND LOCATIONS:
Overall Officials: Harold Lau, MD, Principal Investigator — Tom Baker Cancer Centre